CLINICAL TRIAL: NCT04619160
Title: Influence of Propofol Versus Sevoflurane on Surgical Conditions During Functional Endoscopic Sinus Surgery
Brief Title: Propofol Versus Sevoflurane During FESS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Algemeen Ziekenhuis Maria Middelares (Other)
Responsible Party: Principal Investigator, Dr. Alain Kalmar, MD, PhD, Staff Anesthesist, Algemeen Ziekenhuis Maria Middelares
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MMS.2019.043
Record Dates: First submitted 2020-10-28; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Sinus Infection Chronic
Keywords: haemodynamic; peripheral blood flow; FESS
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The surgeon and participant are blinded for randomization. The anesthesiologist is unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol (Active Comparator)
  Interventions: Drug: Propofol
- sevoflurane (Active Comparator)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — TCI 4 µg/mL start until BIS-value of 50
  Arms: propofol
Drug: Sevoflurane — start 1 MAC, until BIS-value of 50
  Arms: sevoflurane

SUMMARY:
Good surgical conditions are crucial for an optimal surgery result and safe procedure. Minimal blood loss in the surgical field is one of the most important conditions to maintain a good visualization, especially in surgeries with a small surgical field such as a FESS (functional endoscopic sinus surgery). The perioperative blood loss is determined by the main arterial and venous pressure, the local pressure and the capillary vascular filling pressure.

It has been proposed that propofol is a venodilator, which increases the blood flow, but decreases the capillary pressure. On the contrary, sevoflurane might act mainly on the arterioles, which causes an increase in the capillary pressure. In a previous study it has been demonstrated that despite blood pressure maintenance, propofol causes less bleeding during spinal surgery than sevoflurane.

The main aim of this study was to compare both anaesthetics on the perioperative bleeding and haemodynamics during FESS. Secondary, the postoperative nausea, vomiting, pain scores, surgery duration and length of stay at the post-anesthesia care unit will be evaluated.

DETAILED DESCRIPTION:
2 X 30 patients which are planned for FESS surgery are randomized in a sevoflurane group or propofol group.

All patients will be induced with propofol (target-controlled infusion (TCI) 4 µg/mL) and remifentanil (TCI 4 ng/mL) and receive a multimodal intravenous analgesia.

Patients in the propofol group will receive further intravenous propofol until a bispectral index (BIS) value of 50 is reached.

The intravenous drip of propofol will be stopped after induction in the sevoflurane group and patients will receive sevoflurane as inhalation anaesthetic (1 MAC) until a BIS-value of 50. The surgeon will be blinded for patient allocation.

The surgical conditions will be graded postoperatively by the surgeon who performed the operation using the validated Boezaart grading scale. The endoscopic images will be evaluated in addition by 3 blinded surgeons using this same scale.

Besides the surgical conditions, haemodynamic parameters, nausea and vomiting scores (PONV), Visual Analogue Score (VAS), surgery duration, length of stay at the post-anesthesia care unit and postoperative analgesia and anti-emetics are registered.

ELIGIBILITY:
Inclusion Criteria:

* patient planned for FESS surgery

Exclusion Criteria:

* patients which receive anticoagulants
* patients which have coagulation disorders
* patients with high bleeding risk
* patients with arterial hypertension
* other decided by surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Boezaart surgical grading scale | during surgery
  Evaluation of surgical conditions by determination of the validated Boezaart surgical grading scale. Score 0 (no bleeding) to 5 (severe bleeding) The scale will be determined by the operating surgeon and 3 independent surgeons based on an endoscopic video recording.

SECONDARY OUTCOMES:
Surgery duration | Immediately after surgery
  Length of surgery in minutes
Arterial blood pressure | During surgery
  Mean Arterial Blood Pressure (in mmHg)
Length of stay on the PACU | From arrival on the PACU until achievement of the PACU discharge criteria
  number of minutes on the PACU
Postoperative pain scores | in the first 48 hours after surgery
  Postoperative Visual Analogue scores
PONV scores | In the first 48 hours after surgery
  Postoperative nausea/vomiting scores

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, MD, PhD, MSc, Principal Investigator — Maria Middelares Hospital
Locations (1):
- General Hospital Maria Middelares, Ghent, Oost-Vlaanderen, Belgium